CLINICAL TRIAL: NCT03229512
Title: An Open Label, Pilot Study Evaluating the Effect of Topical Sildenafil as Pre-Treatment for Hand-Foot Skin Reaction
Brief Title: Topical Sildenafil as Pre-Treatment for Hand-Foot Skin Reaction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Nam Choi, MD, Chief of Division of Oncodermatology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JNC052716
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hand Foot Skin Reaction
Keywords: Hand Foot Skin Reaction; Sildenafil
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Topical 1% Sildenafil Cream
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Topical 1% Sildenafil Cream
  Other Names: Sildenafil citrate; Viagra

SUMMARY:
Skin toxicities are a major complication to cancer therapies. They can be painful and limit the amount of drug that can be received by cancer patients, preventing the patients from receiving optimal doses of drug. One such cutaneous toxicity, hand-foot skin reaction (HFSR), is caused by next generation targeted agents that are in routine use for the treatment of kidney and liver cancer. HFSR is characterized by swelling, redness, and pain of the palms and soles, in addition to the development of painful or thickened callus-like plaques with fissures in areas of friction and pressure. The investigators have identified a topical skin-directed therapy, 1% topical sildenafil cream, that the investigators believe will be useful in preventing and ameliorating this painful, skin side effect associated with the targeted agents sorafenib and sunitinib. This project proposal aims to conduct an open-label pilot study to assess whether pre-medication with this cream can be an effective way of preventing or decreasing the severity of hand-foot skin reaction, improving their quality of life on therapy and enabling the patients to receive optimal amounts of their anti-cancer drug.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of topical sildenafil as a pre-treatment regimen for HFSR in patients naïve to anti-cancer therapy who will be initiated on treatment with sorafenib or sunitinib. The study endpoint will be the onset and calculated incidence of any grade of HFSR. Skin toxicity grading per National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 will be performed by the investigator at each visit (every 2 weeks) until the end of the study (12 weeks total).

This study aims to:

1. Determine whether HFSR can be prevented with topical sildenafil as pre-treatment.
2. Determine whether topical sildenafil can reduce the incidence of HFSR in patients treated with sorafenib or sunitinib.
3. Determine whether topical sildenafil can delay the onset of HFSR.
4. Determine whether topical sildenafil can reduce the severity of skin lesions if HFSR does occur.

Patient Eligibility:

The target population for this study is patients with clinically-diagnosed cancer who will be treated with sorafenib or sunitinib. A total of 20 subjects will be needed for this trial. There is no placebo group for this study. Subjects must meet all of the inclusion criteria and none of the exclusion criteria to be registered to the study.

Data Collection:

Patients will be instructed to apply the treatment cream to both hands and both feet twice a day for 12 weeks. After the initial visit to enroll and obtain consent, patient assessment will occur in clinic every 2 weeks. At each clinic visit, a skin toxicity grading per NCI-CTCAE v4.03 will be performed, any visual skin changes will be documented with photography, treatment cream will be refilled, and patient medication diaries will be reviewed. A follow up visit will occur within 30 days of the last study treatment. In addition, the investigators will collect information to ensure compliance with drug therapy (in the form of a subject medication diary).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of cancer that are within ± 3 days of initiating treatment with sorafenib or sunitinib. Patients treated with a combination regimen that includes sorafenib or sunitinib are eligible.
* Patients must be age ≥ 18 years.
* Patients must exhibit an ECOG performance status of 0 to 2.
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (e.g., hormonal contraceptives such as birth control pills, patch, intrauterine device; barrier contraception such as male/female condoms, diaphragm; male partner with vasectomy; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy or has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
* FOCBP must have a negative urine or serum pregnancy test within 7 days prior to registration on study.
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration in the study.

Exclusion Criteria:

* Patients with a prior diagnosis of hand-foot skin reaction are not eligible.
* Patients who have had other chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are not eligible.
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to sildenafil or phosphodiesterase-5 (PDE5) inhibitors such as vardenafil (Levitra) and tadalafil (Cialis) are not eligible.
* Patients may not be receiving any other investigational agents. Note: it is acceptable to be on combination therapy including either sorafenib and/or sunitinib.
* Patients must not be using topical steroids (e.g., hydrocortisone). Topical over-the-counter antibiotics (e.g., Neosporin) and skin protectants (e.g., Vaseline, Aquaphor) for local skin fissures on hands and feet are allowed. Patients are allowed to use topical medications on other body parts, besides the hands and feet, but must use qtips or gloves for application.
* Patients taking nitrates (e.g., nitroglycerin, isosorbide mononitrate, isosorbide dinitrate) and/or alpha blockers (e.g., tamsulosin, prazosin, afluzosin, silodosin) are not eligible.
* Patients taking Viagra must have a 1 day washout period prior to treatment. Note: patients must agree to discontinue Viagra while on study treatment.
* Female patients who are pregnant or nursing are not eligible.
* Patients must not have any condition or situation which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study.
* Patients who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Evidence of hand-foot skin reaction | Within 12 weeks of start of study
  The primary outcome measure is the onset and calculated incidence of any grade of hand-foot skin reaction during the 12-week study period.

SECONDARY OUTCOMES:
Adverse events due to 1% sildenafil cream | Within 12 weeks of start of study
  Safety endpoints will include number, frequency and severity of adverse events noted by significant changes upon physical examination or vital sign measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Choi, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Department of Dermatology, Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JN. Chemotherapy-induced iatrogenic injury of skin: new drugs and new concepts. Clin Dermatol. 2011 Nov-Dec;29(6):587-601. doi: 10.1016/j.clindermatol.2011.08.032. PMID 22014981
- [Background] Lacouture ME, Wu S, Robert C, Atkins MB, Kong HH, Guitart J, Garbe C, Hauschild A, Puzanov I, Alexandrescu DT, Anderson RT, Wood L, Dutcher JP. Evolving strategies for the management of hand-foot skin reaction associated with the multitargeted kinase inhibitors sorafenib and sunitinib. Oncologist. 2008 Sep;13(9):1001-11. doi: 10.1634/theoncologist.2008-0131. Epub 2008 Sep 8. PMID 18779536
- [Background] Meadows KL, Rushing C, Honeycutt W, Latta K, Howard L, Arrowood CA, Niedzwiecki D, Hurwitz HI. Treatment of palmar-plantar erythrodysesthesia (PPE) with topical sildenafil: a pilot study. Support Care Cancer. 2015 May;23(5):1311-9. doi: 10.1007/s00520-014-2465-z. Epub 2014 Oct 24. PMID 25341548